CLINICAL TRIAL: NCT06816004
Title: Noninvasive Vagal Nerve Stimulation for the Management of Symptoms Experienced in Multiple Sclerosis (VANISH-MS): An Open-Label Home-Based Study of taVNS and tcVNS Compared to tDCS
Brief Title: Noninvasive Vagal Nerve Stimulation
Acronym: VANISH-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-01628
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: VNS; tDCS; Vagus Nerve Stimulation; Neuromodulation; Multiple Sclerosis; Home-Based
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Active DLPFC tDCS (Active Comparator): 20 daily 20-minute sessions of active tDCS.
  Interventions: Device: Remotely Supervised Transcranial Direct Current Stimulation (RS - tDCS)
- Active taVNS (Experimental): 20 daily 60-minute sessions of active taVNS.
  Interventions: Device: Remotely Supervised Transcutaneous Auricular Vagus Nerve Stimulation (RS - taVNS)
- Active tcVNS (Experimental): 20 daily 20-minute sessions of active tcVNS.
  Interventions: Device: Remotely Supervised Transcutaneous Cervical Vagus Nerve Stimulation (RS - tcVNS)

INTERVENTIONS:
Device: Remotely Supervised Transcranial Direct Current Stimulation (RS - tDCS) — tDCS is a noninvasive brain stimulation device that modulates brain activity delivering a low-intensity electrical current.
  Arms: Active DLPFC tDCS
Device: Remotely Supervised Transcutaneous Auricular Vagus Nerve Stimulation (RS - taVNS) — taVNS is a noninvasive peripheral nerve stimulation device that modulates vagus nerve activity delivering a low-intensity electrical current (< 5mA) through hydrogel electrodes to the left auricular branch of the vagus nerve.
  Arms: Active taVNS
Device: Remotely Supervised Transcutaneous Cervical Vagus Nerve Stimulation (RS - tcVNS) — tcVNS is a noninvasive peripheral nerve stimulation device that modulates vagus nerve activity delivering a low-intensity electrical current (< 5mA) through cervical hydrogel electrodes to the left cervical branch of the vagus nerve.
  Arms: Active tcVNS

SUMMARY:
Growing evidence suggests that vagal nerve stimulation (VNS) may be novel and effective in the management of the symptom burden of multiple sclerosis (MS) potentially by reducing inflammation and emotional distress, therefore improving overall well-being.

We will complete a pilot study comparing transcutaneous auricular vagus nerve stimulation (taVNS) and transcutaneous cervical vagus nerve stimulation (tcVNS) to a standard intervention of dorsolateral prefrontal cortex (DLPFC) transcranial direct current stimulation (tDCS) as an active control. The primary outcome will be feasibility and the preliminary efficacy data concerning self-reported symptom reduction to inform the design of an intervention, and estimated power needed to complete a larger sham-controlled RCT. We will also measure heart rate variability (HRV), an easily obtained biomarker of vagus nerve stimulation (VNS), in correspondence to intervention response.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 25-65 years (inclusive)
* Definite diagnosis of MS or related demyelinating disorders (e.g., Neuromyelitis Optica or NMO)
* Stable high efficacy DMT ≥ 6 months before enrollment and throughout the trial
* PDDS score ≤ 6 (established to be able to complete procedures)
* SymptoMScreen Score ≥12
* WRAT-5 ≥85
* SDMT z-score > -3.0
* K10 < 35
* Stable disease activity, defined as being more than 1 month after a clinical relapse or confirmed radiologic disease activity, or more than 1 month after steroid treatment
* Ability to use mobile devices

Exclusion Criteria:

* Primary neurologic disorder other than MS and related demyelinating disorders like NMO (e.g., stroke, Parkinson's disease, spinal cord injury, intracranial mass, traumatic brain injury (TBI), epilepsy, mild cognitive impairment (MCI), or dementia), psychiatric disorders or major medical disorders (e.g., history of myocardial infarction, diabetes, thyroid disease, arrhythmia, atrial fibrillation)
* Diagnosis of Postural Orthostatic Tachycardia Syndrome (POTS)
* History of vagus nerve surgery/vagotomy
* History of diagnosed cardiovascular disease, a heart transplant, presence of permanent pacemaker implant or Left Ventricular Assist Device
* Use of certain medications that can affect heart rate variability, such as beta-blockers, calcium channel blockers, and cardiac glycosides
* Use of SP1 inhibitor medications such as Fingolimod, Siponimod, Ozanimod, and Ponesimod
* Nicotine use in the past 6 months (smoking/vaping)
* Pregnant or planning pregnancy during the study period or breastfeeding
* Seizure disorder or recent (<5 years) seizure history
* Active ear infections or ear pathology
* Current presence of implanted vagus nerve stimulator or any other active implanted electronic devices (e.g., pacemaker, defibrillators, cochlear implants, DBS, iVNS, etc.)
* Presence of metal objects in the head/neck
* Any skin disorder or skin sensitive area near stimulation locations
* BMI ≥ 35

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Complete Home-Based taVNS or tcVNS Sessions | Up to Week 4 (End of Intervention)
  Assessed among participants in the taVNS or tcVNS arms only.

SECONDARY OUTCOMES:
Change in SymptoMScreen Score | Baseline, Week 4 (End of Intervention)
  SymptoMScreen is a self-report tool to assess overall symptom burden.
Change in Multiple Sclerosis Impact Scale (MSIS-29) Score | Baseline, Week 4 (End of Intervention)
  12-item self-report scale to assess symptom burden regarding neurological domains and the psychological impact of MS. Each item is rated on a 7-point Likert scale from 0 to 6. The item responses are summed to calculate a total score ranging from 0 to 72, with a higher score indicating more severe symptom limitations
Change in Memorial Symptom Assessment Scale (MSAS) Score | Baseline, Week 4 (End of Intervention)
  32-item symptom self-report rating scale to better understand the symptom severity, symptom frequency, and distress from common symptoms. The total MSAS score is the average of the symptom scores for all 32 symptoms and ranges from 0 to 4. Higher scores indicate greater impact from symptoms.
Change in Kessler Psychological Distress Scale (K10) Score | Baseline, Week 4 (End of Intervention)
  10-item questionnaire to assess psychological distress over a recent period of the past 4 weeks focusing on anxiety and depressive symptoms. Each item is rated on a 5-point Likert scale from 1-5. The total score is the sum of responses and ranges from 10-50; higher scores indicate more severe mental disorder.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance - Short Form Score | Baseline, Week 4 (End of Intervention)
  8-item qualitative self-report questionnaire regarding functions of sleep and wakefulness such as perceived sleep quality, sleep depth, and restfulness after sleep in the past 7 days. Each item is rated on a scale from 1-5. The total score is the sum of responses and ranges from 8-40; a higher score indicates more severe sleep disturbances.
Change in PROMIS Fatigue - Short Form 7a Score | Baseline, Week 4 (End of Intervention)
  7-item self-report tool assessing fatigue severity and impact. Each item is rated on a scale from 1-5. The total score is the sum of responses and ranges from 7-35; higher scores indicate greater fatigue.
Change in PROMIS Pain Intensity - Short Form 3a Score | Baseline, Week 4 (End of Intervention)
  3-item tool to evaluate quantitative participant experiences of pain intensity both over the past 7 days and at the time of completing the self-report assessment. Each item is rated on a scale from 1-5. The total score is the sum of responses and ranges from 3-15; higher scores indicate greater pain intensity.
Change in General Anxiety Disorder (GAD-7) Score | Baseline, Week 4 (End of Intervention)
  7-item self-report questionnaire to screen for generalized anxiety in addition to assessing severity of anxiety symptoms. Each item is rated on a scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-21; higher scores indicate more prevalent symptoms of anxiety.
Change in Composite Autonomic Symptom Score-31 (COMPASS-31) Score | Baseline, Week 4 (End of Intervention)
  31-item scale measuring autonomic symptoms in six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor functions. A total score from 0-100 is generated from the item responses; higher scores indicate more severe autonomic dysfunction.
Change in Patient Health Questionnaire (PHQ-9) Score | Baseline, Week 4 (End of Intervention)
  9-item self-report questionnaire to screen for depressive disorder and furthermore, severity. Each item is rated on a scale from 0 (not at all) to 3 (nearly every day). The total score is the sum of responses and ranges from 0-27; higher scores indicate greater severity of depressive symptoms.
Change in Nine-Hole Peg Test (9HPT) Score | Baseline, Week 4 (End of Intervention)
  Assessment of manual dexterity and fine motor coordination in people with MS, using both dominant and non-dominant hands. The score is measured by the number of seconds it takes for a person to place and remove nine pegs from a pegboard, with a lower score (in seconds) indicating better dexterity and faster completion time.
Change in Heart Rate Variability (HRV) | Baseline, Week 4 (End of Intervention)
  Assessed using the Chest Strap Polar H10 HR sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.